CLINICAL TRIAL: NCT02068495
Title: Unisia Combination Tablets LD, HD Special Drug Use Surveillance "Hypertension: Long-Term Use"
Brief Title: Candesartan Cilexetil/Amlodipine Besilate Combination Tablets LD, HD Special Drug Use Surveillance "Hypertension: Long-Term Use"
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 119-011; JapicCTI-132390 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2014-02-19; First posted 2014-02-21 (Estimated); Results first posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Hypertension
Keywords: Drug therapy
MeSH Terms: conditions — Hypertension | interventions — candesartan cilexetil; Amlodipine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Candesartan cilexetil/Amlodipine besilate: 8 milligram (mg)/2.5 mg or 8 mg/5 mg, orally, once daily
  Interventions: Drug: Candesartan cilexetil/Amlodipine besilate

INTERVENTIONS:
Drug: Candesartan cilexetil/Amlodipine besilate — Candesartan cilexetil/Amlodipine besilate tablets
  Other Names: Unisia Combination Tablets

SUMMARY:
The purpose of this survey is to investigate the safety and efficacy of long-term use of candesartan cilexetil/amlodipine besilate combination tablets (Unisia Combination Tablets) low dose (LD), high dose (HD) in participants with hypertension in the normal clinical setting.

DETAILED DESCRIPTION:
This special drug use surveillance was designed to investigate the safety and efficacy of long-term use of candesartan cilexetil/amlodipine besilate combination tablets (Unisia Combination Tablets) in participants with hypertension in the routine clinical setting.

The usual adult dosage is one tablet (8 mg/2.5 mg or 8 mg/5 mg as candesartan cilexetil/amlodipine besilate) administered orally once daily.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with hypertension

Exclusion Criteria:

1. Participants in whom Candesartan cilexetil/Amlodipine besilate is contraindicated [Contraindications]
2. Participants with a history of hypersensitivity to the ingredients of Candesartan cilexetil/Amlodipine besilate or any other dihydropyridine formulations
3. Women who are pregnant or of child-bearing potential

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hypertension
Sampling Method: Non-Probability Sample
Enrollment: 3409 (Actual)
Dates: Start 2010-06-15 (Actual); Primary Completion 2013-05-31 (Actual); Study Completion 2013-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 579 investigative sites in Japan, from 15 June 2010 to 31 May 2013.
Pre-assignment Details: Participants with a historical diagnosis of hypertension were enrolled to receive Candesartan cilexetil/Amlodipine 8 milligram (mg)/2.5 mg - 8 mg/5 mg combination tablet, orally, once daily for up to 12 months.
Groups:
- Candesartan Cilexetil/Amlodipine: Candesartan cilexetil/Amlodipine 8 mg/2.5 mg - 8 mg/5 mg combination tablet, orally, once daily for up to 12 months in participants based upon the disease severity. Participants received interventions as part of routine medical care.
Period: Overall Study
Arm/Group | Candesartan Cilexetil/Amlodipine
Started | 3409
Completed | 3300
Not Completed | 109
Not completed — Case Report Forms Uncollected | 60
Not completed — Protocol Deviation | 49

BASELINE CHARACTERISTICS:
Population: The safety analysis set was defined as all participants who were enrolled and completed the study.
Arm/Group | Candesartan Cilexetil/Amlodipine
Number analyzed (Participants) | 3300
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.8 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1692
  Male | 1608
Region of Enrollment [Number; unit: Participants]
  Japan | 3300
Duration of Hypertension [Mean (Standard Deviation); unit: Years] — Mean Duration between start of study and first time of diagnosis of hypertension was reported.
  Years | 6.29 (6.57)
Healthcare Category [Count of Participants; unit: Participants] — Participants were categorized as outpatient, inpatient, and outpatient and inpatient (participants who were both outpatient and inpatient throughout study).
  Participants
    Outpatient | 3222 (3.83)
    Inpatient | 8
    Outpatient and Inpatient | 70
Non Breast-Feeding Females [Count of Participants; unit: Participants] — Population: This baseline characteristic was analyzed only in female participants.
  Participants
    number analyzed (Participants) | 1692
    (all) | 1692
History of Allergy [Count of Participants; unit: Participants]
  Had No Presence of History of Allergy | 2872
  Had Presence of History of Allergy | 222
  Unknown | 206
Medical Complications [Count of Participants; unit: Participants] — Complications defined as a disease or a health condition for each participant at the start of study. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications. Other complications included all complications except for those mentioned above.
  Participants
    Had No Presence of Medical Complications | 791
    Had Presence of Medical Complications | 2509
Medical History [Count of Participants; unit: Participants]
  Had No Presence of Medical History | 2567
  Had Presence of Medial History | 630
  Unknown | 103
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 60.43 (13.04)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index = weight (kg)/[height (m)^2]
  kg/m^2 | 24.14 (3.83)
Waist Circumference [Mean (Standard Deviation); unit: centimeter (cm)]] | 86.47 (9.85)
Drinking Habits [Count of Participants; unit: Participants]
  Never Drank | 1707
  Current Drinker | 942
  Ex-Drinker | 200
  Unknown | 451
Smoking Classification [Count of Participants; unit: Participants]
  Never Smoked | 2066
  Current Smoker | 402
  Ex-Smoker | 383
  Unknown | 449
Use of Antihypertensive Drug Prior to the Start of the Study Drug [Count of Participants; unit: Participants]
  Had Not Used Antihypertensive Drug | 200
  Had Used Antihypertensive Drug | 3100

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experience at Least One Adverse Events
Time Frame: Up to 12 Months
Population: The safety analysis set was defined as all participants who were enrolled and completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Candesartan Cilexetil/Amlodipine
Number analyzed (Participants) | 3300
Participants | 286

2. Primary Outcome: Number of Participants Who Experience at Least One Adverse Drug Reactions (ADRs)
Description: ADRs are defined as adverse events (AEs) which are in the investigator's opinion of causal relationship to the study treatment. AEs are defined as any unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product reported from the first dose of study drug to the last dose of study drug.
Time Frame: Up to 12 Months
Population: The safety analysis set was defined as all participants who were enrolled and completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Candesartan Cilexetil/Amlodipine
Number analyzed (Participants) | 3300
Participants | 85

3. Secondary Outcome: Changes From Baseline in Systolic Blood Pressure (SBP) at Final Assessment
Description: Reported data are changes in SBP from baseline at final assessment (up to 12 months).
Time Frame: Baseline and final assessment (up to 12 Months)
Population: The efficacy assessment population was defined as participants who completed the study and had efficacy data at baseline and post-baseline time points available. Here 'Number of Participants Analyzed' is number of participants analyzed at the given populations.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Candesartan Cilexetil/Amlodipine
Number analyzed (Participants) | 3246
mmHg | -14.6 (19.6)

4. Secondary Outcome: Changes From Baseline in Diastolic Blood Pressure (DBP) at Final Assessment
Description: Reported data are changes in DBP from baseline at final assessment (up to 12 months).
Time Frame: Baseline and final assessment (up to 12 Months)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Candesartan Cilexetil/Amlodipine
Number analyzed (Participants) | 3246
mmHg | -7.2 (12.3)

5. Secondary Outcome: Changes From Baseline in Pulse Rate at Final Assessment
Description: Reported data are changes in Pulse Rate from baseline at final assessment (up to 12 months).
Time Frame: Baseline and final assessment (up to 12 Months)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Candesartan Cilexetil/Amlodipine
Number analyzed (Participants) | 2259
Beats per minute | -1.2 (10.2)

6. Secondary Outcome: Percentage of Participants Who Meet Targeted Blood Pressure Level at Baseline and Final Assessment
Description: Reported data are percentage of participants who meet targeted blood pressure level at baseline and final assessment in analysis population. Targeted blood pressure level of SBP/DBP was less than 140/90 mmHg.
Time Frame: Baseline and final assessment (up to 12 Months)
Population: The efficacy assessment population was defined as participants who completed the study and had efficacy data at baseline and post-baseline time points available. Here 'Number of Participants Analyzed' is number of participants analyzed at the given time point.
Measure: Number; unit: Percentage of Participants
Arm/Group | Candesartan Cilexetil/Amlodipine
Number analyzed (Participants) | 3246
Percentage of Participants
  Baseline | 28.5
  Final Assessment | 66.9

ADVERSE EVENTS:
Time Frame: Up to 12 Months
Description: At each visit the investigator had to document any occurrence of AEs and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Participants may be represented in more than 1 category.
Arm/Group | Candesartan Cilexetil/Amlodipine
Serious Adverse Events (participants affected / at risk) | 63/3300
Other Adverse Events (participants affected / at risk) | 97/3300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Candesartan Cilexetil/Amlodipine (N=3300)
Peritonitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 6
Pyelonephritis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Infectious pleural effusion (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Liver carcinoma ruptured (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Marasmus (Metabolism and nutrition disorders) | 3
Completed suicide (Psychiatric disorders) | 1
Cerebral infarction (Nervous system disorders) | 3
Dementia Alzheimer's type (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Motor neurone disease (Nervous system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Atrioventricular block complete (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 3
Cardiac failure acute (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Myocardial ischaemial (Cardiac disorders) | 1
Sick sinus syndrome (Cardiac disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Diverticulitis intestinal haemorrhagic (Gastrointestinal disorders) | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Hepatic Failure (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Renal artery stenosis (Renal and urinary disorders) | 1
Renal disorder (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Renal failure chronic (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Death (General disorders) | 1 — The reasons of events are not determined because assessment findings were insufficient to specify the reason.
Oedema peripheral (General disorders) | 1
Blood creatinine increased (Investigations) | 1
Blood pressure decreased (Investigations) | 1
Blood urea increased (Investigations) | 1
Fall (Injury, poisoning and procedural complications) | 2
Humerus fracture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 4
Thermal burn (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Pubis fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 0.3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Candesartan Cilexetil/Amlodipine (N=3300)
Dizziness (Nervous system disorders) | 15
Hepatic function abnormal (Hepatobiliary disorders) | 18
Blood creatinine increased (Investigations) | 12
Blood pressure decreased (Investigations) | 21
Blood urea increased (Investigations) | 17
Gamma-glutamyltransferase increased (Investigations) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.